CLINICAL TRIAL: NCT07228221
Title: iStent Infinite and iDose TR for Management of Moderate to Severe Primary Open Angle Glaucoma Are a Safe and Effective Alternative to Filtering Surgery for IOP Reduction in Patients With Medically Uncontrolled Glaucoma. (POAG)
Brief Title: Standalone iStent Infinite and iDose TR for Management of Moderate to Severe Open Angle Glaucoma
Acronym: POAG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jonathon Myers (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jonathon Myers, Co-Investigator, Wills Eye
Organization: Wills Eye (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WEH IRB #2025-51
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Open Angle Glaucoma; Pigmentary Glaucoma; Pseudoexfoliation Glaucoma
Keywords: POAG; PG; PXG
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Intervention Model Description: Each patient will have surgery using the iStent infinite Trabecular Micro-bypass model iS3 and the iDose TR (Travoprost Intracameral Implant) 75mcg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surgery for patients with medically uncontrolled POAG (Experimental): surgery using combined minimally invasive surgical iStent infinite trabecular micro-bypass systme model iS3 and drug depot iDose TR (Travoprost Intracameral Implant) 75mcg
  Interventions: Device: iStent infinite trabecular micro-bypass system model iS3; Drug: iDose TR (Travoprost intracameral Implant) 75mcg

INTERVENTIONS:
Device: iStent infinite trabecular micro-bypass system model iS3 — surgery perfomed using the iStent infinite trabecular micro-bypass system model iS3
Drug: iDose TR (Travoprost intracameral Implant) 75mcg — surgery performed using the iDose TR (Travoprost intracameral Implant) 75mcg

SUMMARY:
The Investigators will investigate the efficacy of combining the standalone iStent infinite and iDose that are minimally invasive surgical and drug depot options are a safe and effective alternative to filtering surgery for intraocuar pressure reduction in patients with medically uncontrolled open angle glaucoma.

DETAILED DESCRIPTION:
The Investigators will assess the mean intraocular pressure change from baseline, the change in the number of medications from baseline, the proportion of patients needing additional incisional surgery, and the incidence of adverse events. The Investigators hypothesize that patients receiving the combined standalone iStent infinite and iDose will experience a safe and significant reduction in mean intraocular pressure and number of medications during the study time period.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe open angle glaucoma (including POAG, PG, and PXG)
* Open angle configuration (Shaffer grade ≥ 3), normal angle anatomy9
* Visual acuity HM or better
* VF MD -6dB or worse
* Failed medical therapy and/or laser treatment
* Incisional glaucoma surgery contemplated as next intervention
* Phakic or pseudophakic

Exclusion Criteria:

* Traumatic, uveitic, neovascular glaucoma, or angle closure glaucoma
* Previous incisional glaucoma surgery
* ALT; History of iridotomy, SLT, or micropulse laser trabeculoplasty within the prior 90 days
* Active ocular inflammation or edema, clinically significant corneal dystrophy
* Corneal or other pathology preventing accurate Goldmann applanation tonometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2031-08-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
IOP reduction from baseline | Diurnal IOP reduction from baseline at 12 months
  a logistic regression model will be used for the imputation of missing values, using the 12-month performance outcome as dependent variable, and sex, race, age, baseline IOP, number of IOP-lowering medications used at baseline, last IOP and number of medications at the 6-month visit or later as explanatory variables.

CONTACTS AND LOCATIONS:
Overall Officials: Dilru Amarasekera, MD, Principal Investigator — Wills Eye Hospital Glaucoma Research
Locations (1):
- Wills Eye Hosital Glaucoma Dept., Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, Statistical Analysis Plan (SAP), informed Consent Form, and deidentified participant and group data will be kept on file at Wills Eye Hospital for 7 years. Researchers can request this data by email to glaucoma@willseye.org with a description of their planned use.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: This is a 5 year study with anticipated completion of enrollment and data December 2031.
Access Criteria: Researchers can request the study protocol, Statistical Analysis Plan (SAP), informed Consent Form, and deidentified participant and group data with a description of their planned use
URL: https://www.gresearch@willseye.org